CLINICAL TRIAL: NCT04948853
Title: Improving Employment Outcomes for Probationers With Mental Illnesses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: U.S. Department of Justice (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 21-0972; 2019-MO-BX-0022 (Other Grant/Funding Number: Department of Justice)
Record Dates: First submitted 2021-06-23; First posted 2021-07-02 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Mental Disorders, Severe
Keywords: probation; employment
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Intervention Model Description: Randomized control trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment as usual (No Intervention): Treatment as usual, with respect to employment, for individuals on probation typically entails the probation officer informing the probationer that probationer is responsible for obtaining employment or could entail a referral from a probation officer to an employment or job assistance service, such as vocational rehabilitation. The probationer is responsible for follow up with that service.
- Intervention - Individual Placement Support-Supported Employment (Experimental): Subjects in this condition will receive services from a 1.5 FTE IPS-SE team that will work to provide one-on-one person-centered services to help obtain employment, including but not limited to career profiling, resume assistance, job placement, training and other activities.
  Interventions: Behavioral: Individual Placement Support - Supported Employment

INTERVENTIONS:
Behavioral: Individual Placement Support - Supported Employment — Individual, person-centered intervention designed to help individuals living with mental illnesses obtain and sustain meaningful employment. This is an evidence-based practice for individuals with severe mental illnesses.
  Arms: Intervention - Individual Placement Support-Supported Employment

SUMMARY:
Employment is a key protective factor against recidivism; however, the lack of job opportunities keeps justice-involved mentally ill individuals, especially young adults of color, unemployed and at risk for future justice involvement. To address these issues and grow the evidence for evidence-based practices for justice-involved adults with mental illnesses, the investigators will study the implementation and outcomes of individual placement support-supported employment (IPS-SE) combined with specialty mental health probation (SMHP) for probationers with mental illnesses.

DETAILED DESCRIPTION:
The large and growing number of individuals with mental illnesses who are on probation have a difficult time accessing housing, employment, and health and mental health care, which is especially concerning for young adults aged 19-25 who make up just 10% of the population but 26% of those on probation. Employment is a key protective factor against recidivism; however, the lack of job opportunities keeps justice-involved mentally ill individuals, especially young adults of color, unemployed and at risk for future justice involvement. Without access to evidence-based supported employment interventions, economic inequality and poverty among justice-involved young adults with mental illnesses will remain unchanged.

To this end, an experienced multidisciplinary team will study the implementation and outcomes of individual placement support-supported employment (IPS-SE) combined with specialty mental health probation (SMHP) for probationers with mental illnesses. The investigators' long-term goal is to develop the evidence for interventions designed to improve employment outcomes among justice-involved individuals who have mental illnesses and conduct translational research with broad application to justice-involved individuals living with mental illnesses. The investigators will pursue the following specific aims:

Aim 1: Examine the barriers and facilitators to implementing IPS-SE in a probation setting. The investigators will use qualitative methods and semi-structured interviews with key stakeholders involved in the implementation of SMHP+IPS-SE to understand how IPS-SE can be embedded successfully in a probation setting.

Aim 2: Conduct a randomized trial to examine the impact of the SMHP+IPS-SE on employment and annual income for probationers with mental illnesses. The investigators will randomly assign 120 individuals to receive SMHP + treatment as usual (TAU) or SMHP+IPS-SE. The research team will test the following hypothesis - H1: SMHP+IPS-SE recipients will be more likely to obtain and sustain employment compared to SMHP+TAU recipients.

The expected outcomes include: (1) an understanding of the implementation barriers and facilitators associated with providing IPS-SE in a probation setting; (2) an understanding of how IPS-SE needs to be adapted for probationers with mental illnesses; and (3) evidence that SMHP+IPS-SE can improve employment outcomes among justice-involved probationers with mental illnesses. This research has the potential to promote the adoption and dissemination of best practices at the interface of the mental health and criminal justice systems and promises to grow the evidence for interventions that improve employment and reduce economic inequalities among a vulnerable population.

ELIGIBILITY:
Inclusion criteria include:

* on probation and supervised by a SMHP officer;
* aged 18-99;
* interested in obtaining employment; and
* competent to provide informed consent.

Exclusion criteria:

* Does not meet inclusion criteria; and
* Unable/unwilling to provide informed consent

Ages: 19 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Employment, Time 0 | Baseline (Time 0)
  Absence or presence of employment - categorical variable (full-time, part-time, none)
Employment, Time 1 | 3-months (Time 1)
  Absence or presence of employment - categorical variable (full-time, part-time, none)
Employment, Time 2 | 6-months (Time 2)
  Absence or presence of employment - categorical variable (full-time, part-time, none)
Days worked in past 30 days, Time 0 | Baseline (Time 0)
  Number of days worked in last 30 days
Days worked in past 30 days, Time 1 | 3-months (Time 1)
  Number of days worked in last 30 days
Days worked in past 30 days, Time 2 | 6-months (Time 2)
  Number of days worked in last 30 days

SECONDARY OUTCOMES:
Duke-UNC Functional Social Support Questionnaire (FSSQ) | Baseline (Time 0)
  This is an 8-item self-report measure of perceived social support. Scores on the FSSQ range from 8 - 40 with higher scores indicating higher levels of perceived social support.
Duke-UNC Functional Social Support Questionnaire (FSSQ) | 3-months (Time 1)
  This is an 8-item self-report measure of perceived social support. Scores on the FSSQ range from 8 - 40 with higher scores indicating higher levels of perceived social support.
Duke-UNC Functional Social Support Questionnaire (FSSQ) | 6-months (Time 2)
  This is an 8-item self-report measure of perceived social support. Scores on the FSSQ range from 8 - 40 with higher scores indicating higher levels of perceived social support.
Symptom Checklist (SCL-10-R) | Baseline (Time 0)
  This is a 10-item self-report measure of mental health symptom distress. Scores on the SCL-10-R range from 0 - 40 with higher scores indicating higher levels of symptom distress.
Symptom Checklist (SCL-10-R) | 3-months (Time 1)
  This is a 10-item self-report measure of mental health symptom distress. Scores on the SCL-10-R range from 0 - 40 with higher scores indicating higher levels of symptom distress.
Symptom Checklist (SCL-10-R) | 6-months (Time 2)
  This is a 10-item self-report measure of mental health symptom distress. Scores on the SCL-10-R range from 0 - 40 with higher scores indicating higher levels of symptom distress.
Rosenberg Self-Esteem Scale (RSE) | Baseline (Time 0)
  This is a 10-item self-report measure of self-esteem. Scores on the RSE range from 10 - 40 with higher scores indicating greater self-esteem.
Rosenberg Self-Esteem Scale (RSE) | 3-months (Time 1)
  This is a 10-item self-report measure of self-esteem. Scores on the RSE range from 10 - 40 with higher scores indicating greater self-esteem.
Rosenberg Self-Esteem Scale (RSE) | 6-months (Time 2)
  This is a 10-item self-report measure of self-esteem. Scores on the RSE range from 10 - 40 with higher scores indicating greater self-esteem.
Quality of Life (QOL) | Baseline (Time 0)
  This is a 17-item self-report measure of quality of life. Scores on the QOL range from 17 - 68 with higher scores indicating greater quality of life.
Quality of Life (QOL) | 3-months (Time 1)
  This is a 17-item self-report measure of quality of life. Scores on the QOL range from 17 - 68 with higher scores indicating greater quality of life.
Quality of Life (QOL) | 6-months (Time 2)
  This is a 17-item self-report measure of quality of life. Scores on the QOL range from 17 - 68 with higher scores indicating greater quality of life.
Employment Motivation/Readiness (EMR) | Baseline (Time 0)
  This is a 7-item self-report measure of motivation to become employed and readiness to engage with an employment service. Scores on the EMR range from 0 - 70 with higher scores indicating greater motivation and readiness to work.
Employment Motivation/Readiness (EMR) | 3-months (Time 1)
  This is a 7-item self-report measure of motivation to become employed and readiness to engage with an employment service. Scores on the EMR range from 0 - 70 with higher scores indicating greater motivation and readiness to work.
Employment Motivation/Readiness (EMR) | 6-months (Time 2)
  This is a 7-item self-report measure of motivation to become employed and readiness to engage with an employment service. Scores on the EMR range from 0 - 70 with higher scores indicating greater motivation and readiness to work.
Internalized Stigma of Mental Illness (ISMI) | Baseline (Time 0)
  This is a 29-item self-report measure of internalized and socialized stigma of mental illness. Scores on the ISMI range from 29 - 116 with higher scores indicating greater perceived stigma.
Internalized Stigma of Mental Illness (ISMI) | 3-months (Time 1)
  This is a 29-item self-report measure of internalized and socialized stigma of mental illness. Scores on the ISMI range from 29 - 116 with higher scores indicating greater perceived stigma.
Internalized Stigma of Mental Illness (ISMI) | 6-months (Time 2)
  This is a 29-item self-report measure of internalized and socialized stigma of mental illness. Scores on the ISMI range from 29 - 116 with higher scores indicating greater perceived stigma.

CONTACTS AND LOCATIONS:
Overall Officials: Gary S Cuddeback, Ph.D., Principal Investigator — Virginia Commonwealth University; Tonya VanDeinse, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
In the interest of reinforcing open scientific inquiry, data from this study will be made available by the Principal Investigator (PI) as freely as possible while safeguarding the confidentiality and privacy of participants. A final research data set will be prepared containing de-identified data on the ~130 expected participants. A data-sharing agreement will be required and those seeking data access will be required to obtain ethics approval. Researchers with a convincing scientific interest in the data will be eligible to receive the data. The data-sharing agreement will provide for the use of the data only for research and no other purpose, require a plan for the security of the data, forbid the further dissemination of the data without entering into an agreement, and provide a deadline for the completion of analyses and destruction of the data. Data will be made available under the auspices of the PIs by secure file transfer protocols or other secure, industry-approved means.
Time Frame: The data will become available 24 calendar months after completion of the study. The data will be available for up to 5 years.
Access Criteria: Upon request for the data to be shared and evidence of ethics approval, a data-sharing agreement will be required. Researchers with a convincing scientific interest in the data will be eligible to receive the data, without regard for the type of research question.